CLINICAL TRIAL: NCT05045755
Title: The Durability of Protection and Immuno-persistence Study of A Bivalent Human Papillomavirus (Type 16, 18) Recombinant Vaccine (E.Coli) in Healthy Women Aged 18 to 45 Years
Brief Title: The Durability of Protection and Immuno-persistence Study of a Recombinant HPV 16/18 Bivalent Vaccine in Female
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jun Zhang (Other)
Collaborators: Xiamen Innovax Biotech Co., Ltd (Industry); Beijing Wantai Biological Pharmacy Enterprise Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Jun Zhang, Professor, Xiamen University
Organization: Xiamen University (Other)
Other Study IDs: HPV-PRO-003-2
Record Dates: First submitted 2021-07-13; First posted 2021-09-16 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Cervical Intraepithelial Neoplasia; Cervical Cancer; Vaginal Intraepithelial Neoplasia; Vulvar Intraepithelial Neoplasia; Persistent Infection
Keywords: Durability of Protection; Immuno-persistence; Human Papillomavirus 16; Human Papillomavirus 18; vaccine; females
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms; Persistent Infection | interventions — Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vaccine group: Participants in this arm have received 3 doses of HPV 16/18 bivalent vaccine that contains 40μg HPV 16 virus-like particle antigen and 20μg HPV 18 virus-like particle antigen adsorbed in alum-adjuvant.
  Interventions: Biological: Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Escherichia coli)
- Control group: Participants in this arm have received 3 doses of HEV vaccine that contains 30μg HEV virus-like particle antigen adsorbed in alum-adjuvant.

INTERVENTIONS:
Biological: Recombinant Human Papillomavirus Bivalent (Types 16, 18) Vaccine (Escherichia coli) — The bivalent HPV-16/18 vaccine was a mixture of two aluminum hydroxide adjuvant-absorbed recombinant L1 VLPs of HPV-16 and HPV-18 expressed in E. coli. A 0.5 ml dose of the bivalent HPV test vaccine comprised 40 μg of HPV-16 and 20 μg of HPV-18 L1 VLPs absorbed with 208 μg of aluminum adjuvant
  Other Names: There is no other Intervention in this study
  Groups: Vaccine group

SUMMARY:
The primary objective of this study is to evaluate the durability of protection and immuno-persistence of Recombinant Human Papillomavirus Bivalent (Types 16,18) Vaccine administered in females aged 18-45 years.

DETAILED DESCRIPTION:
This is a follow-up study that is based on phase III clinical study of a recombinant human papillomavirus 16/18 bivalent vaccine in females aged 18-45 years (Unique Protocol ID: HPV-PRO-003, Identifiers: NCT01735006). The investigators will recruit people who have participated in phase III clinical study before and to evaluate the durability of protection and immuno-persistence of the bivalent HPV vaccine on 90m and 114m after dose 1.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who participated in the Phase III clinical study of a recombinant human papillomavirus 16/18 bivalent vaccine in females (Unique Protocol ID: HPV-PRO-003, Identifiers: NCT01735006) and received at least one dose;
2. Participants can fully understand the study content and sign an informed consent form；
3. Able to comply with the requests of the study;

Exclusion Criteria:

1. Participants used other HPV vaccine products (including both marketed and unmarketed vaccines) since participating in the Phase III clinical study.
2. According to the investigator's judgment, there might be some medical, psychological, social or occupational factors which might impact on the individual to obey the protocol or sign the informed consent;

Ages: 26 Years to 54 Years | Sex: Female
Age Groups: Adult
Study Population: In Henan Province, participants who participated in the Phase III clinical study of a recombinant human papillomavirus 16/18 bivalent vaccine in females (Unique Protocol ID: HPV-PRO-003, Identifiers: NCT01735006) and received at least one dose
Sampling Method: Non-Probability Sample
Enrollment: 1339 (Estimated)
Dates: Start 2021-04-13 (Actual); Primary Completion 2023-08-10 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects With CIN2+ and/or VIN2+ and/or VaIN2+ Associated With HPV-16 and/or -18 Cervical Infection on 90m and 114m after dose 1 | expected 2-3 years
  To observe the number of Subjects With Histopathologically-confirmed CIN2+ and/or VIN2+ and/or VaIN2+ Associated With HPV-16 and/or -18 Cervical Infection on 90m and 114m after dose 1
Number of Subjects With HPV-16 and/or -18 persistent cervical infection(6-month+ definition) on 90m and 114m after dose 1 | expected 2-3 years
  To detect the HPV16 and HPV18 DNA on the gynecological specimens ( Cervical exfoliated cell specimens and biopsy specimens) collected from the subjects

SECONDARY OUTCOMES:
Anti-HPV16 and anti-HPV18 type-specific IgG antibody level on 90m and 114m after dose 1 | expected 2-3 years
  To detect the anti-HPV 16 and anti-HPV 18 seroconversion rates and geometric mean concentrations on 90m and 114m after dose 1

CONTACTS AND LOCATIONS:
Overall Officials: Ting Wu, Ph. D., Study Chair — Xiamen University
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China